CLINICAL TRIAL: NCT00597402
Title: Avastin in Combination With Radiation and Temozolomide, Followed by Avastin, Temozolomide and Irinotecan for Glioblastoma Multiformes and Gliosarcomas
Brief Title: Avastin in Combination With Radiation (XRT) & Temozolomide, Followed by Avastin, Temozolomide and Irinotecan for Glioblastoma (GBM) and Gliosarcomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Genentech, Inc. (Industry); Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00000458
Record Dates: First submitted 2008-01-10; First posted 2008-01-18 (Estimated); Results first posted 2013-01-18 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-04

CONDITIONS: Glioblastoma; Gliosarcoma; Brain Tumor
Keywords: Avastin; Bevacizumab; Temozolomide; Temodar; Irinotecan; Camptosar; GBM; Glioblastoma Multiforme; Gliosarcoma; Brain tumor; Glioma; New GBM; Newly diagnosed GBM or gliosarcoma malignant brain tumor
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms; Glioma | interventions — Bevacizumab; Temozolomide; Radiotherapy; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Avastin, radiation, temozolomide, and irinotecan (Experimental)
  Interventions: Drug: Avastin; Drug: Temozolomide; Radiation: Radiation Therapy (XRT); Drug: Irinotecan

INTERVENTIONS:
Drug: Avastin — Avastin will be administered 10 mg/kg every other week beginning a minimum of 28 days after last major surgical procedure, open biopsy, or significant traumatic injury. Following completion of XRT, patients will receive treatment that includes 6 cycles of Avastin, beginning a minimum of 14 days after last XRT.
  Other Names: Bevacizumab
Drug: Temozolomide — Daily temozolomide 75 mg/m2/day for 6.5 weeks of radiation treatment. Following completion of XRT, patients will receive treatment including temozolomide 200 mg/m2/day on the 1st 5 days of each 28-day cycle.
  Other Names: Temodar
Radiation: Radiation Therapy (XRT) — Treatment with standard XRT (radiation) for 6.5 weeks.
Drug: Irinotecan — Following completion of XRT, patients will receive 6 cycles of treatment that includes irinotecan. Beginning a minimum of 14 days after last XRT, the irinotecan dose will depend on whether the patient is on enzyme-inducing antiepileptic drugs (EIAED). (EIAED:340 mg/m2 every other week, non-EIAED: 125 mg/m2.)
  Other Names: CPT-11; Camptosar

SUMMARY:
Primary objective: To use overall survival to assess the efficacy of the combination of radiation therapy, temozolomide and Avastin followed by Avastin, temozolomide, and irinotecan in the treatment of grade IV malignant glioma patients following surgical resection.

Secondary objective: To determine the progression-free survival following the combination of radiation therapy, temozolomide and Avastin followed by Avastin, temozolomide, and irinotecan.

Exploratory Objective: To explore the relationship between biomarkers and outcome (overall survival and progression-free survival) among patients with grade IV malignant glioma treated with radiation therapy, temozolomide and Avastin followed by Avastin, temozolomide, and irinotecan.

To describe the toxicity of radiation therapy,temozolomide and Avastin followed by Avastin, temozolomide, and irinotecan.

DETAILED DESCRIPTION:
The standard of care for grade IV gliomas is radiation therapy with daily temozolomide, followed by 6 months of temozolomide. The majority of patients progress and die of their tumor. Many glioma patients are resistant to temozolomide because the tumors have high O(6)-methylguanine-DNA methyltransferase (MGMT), conferring resistance. Irinotecan is synergistic with temozolomide, and the combination may overcome high MGMT. Vascular endothelial growth factor (VEGF) is present on the cell surface and around malignant gliomas. It appears that the presence of vascular endothelial growth factor is a prognostic growth factor with more VEGF expression correlating with a poor prognosis. Monoclonal antibodies to VEGF have inhibited growth of malignant gliomas in a mouse xenograft. Avastin is a humanized monoclonal immunoglobulin G (IGG) 1 antibody that binds to and inhibits the biologic activity of human vascular endothelial growth factor. The combination of Avastin and irinotecan was safe and demonstrated high activity against recurrent malignant gliomas. The combination of Avastin, temozolomide, and irinotecan as the initial therapy may maximize the chance for long-term survival. There are other studies completed or ongoing for newly diagnosed glioblastoma (GBM) patients, including a Radiation Therapy Oncology Group (RTOG) study that added irinotecan to temozolomide following standard radiation therapy and temozolomide, and a University of California, Los Angeles (UCLA) study that added Avastin to standard radiation therapy and temozolomide followed by Avastin and temozolomide.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed diagnosis of World Health Organization (WHO) grade IV primary malignant glioma (glioblastoma multiforme or gliosarcoma). Patients have to be within 4 weeks of the last major surgical procedure.
* Age > 18 years.
* An interval of at least 2 weeks and not > 6 weeks between prior major surgical procedure and study enrollment.
* No prior radiotherapy or chemotherapy for a brain tumor
* Karnofsky ≥ 60 percent.
* Hemoglobin ≥ 9.0 g/deciliter (dl), absolute neutrophil count (ANC) ≥ 1,500 cells/ microliter, platelets ≥ 125,000 cells/microliter.
* Serum creatinine ≤ 1.5 mg/dl, serum serum glutamic-oxaloacetic transaminase (SGOT) and bilirubin ≤ 1.5 times upper limit of normal (ULN).
* For patients on corticosteroids, they must be on a stable or decreasing dose for 1 week prior to entry, and the dose should not be escalated over entry dose level, if clinically possible.
* Signed informed consent approved by the Institutional Review Board
* No evidence of > grade 1 central nervous system (CNS) hemorrhage on the baseline MRI or CT scan.
* If sexually active, patients will take contraceptive measures for the duration of treatment as stated in the informed consent.

Exclusion Criteria:

* Pregnancy or breast feeding.
* Co-medication that may interfere with study results; e.g. immuno-suppressive agents other than corticosteroids.
* Active infection requiring intravenous (IV) antibiotics.
* Prior treatment with radiotherapy or chemotherapy for a brain tumor, irrespective of the grade of the tumor.
* Evidence of > grade 1 CNS hemorrhage on baseline MRI on CT scan.

Avastin-Specific Concerns:

Subjects meeting any of the following criteria are ineligible for study entry:

* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study
* Blood pressure of 150/100 mmHg
* Unstable angina
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infarction within 6 months
* History of stroke within 6 months
* Clinically significant peripheral vascular disease
* Evidence of bleeding diathesis
* Coagulopathy (prothrombin time (PT) or partial thromboplastin time (PTT) >1.5x normal or a history of > three grade 2 or greater hemorrhages)
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to first Avastin infusion during XRT/Temodar or anticipation of need for major surgical procedure during the course of the study
* Minor surgical procedures, fine needle aspirations or core biopsies within 7 days prior to first Avastin infusion during XRT/Temodar
* Pregnant (positive pregnancy test) or lactating
* Urine protein >1.0 + at screening
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to first Avastin infusion during XRT/Temodar
* Serious, non-healing wound, ulcer, or bone fractures.
* Inability to comply with study and/or follow-up procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2007-07; Primary Completion 2011-08 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annick Desjardins, MD, FRCPC, Principal Investigator — Duke Health
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

REFERENCES:
- See also: The Preston Robert Tisch Brain Tumor Center at DUKE — http://www.cancer.duke.edu/btc/

RESULTS

PARTICIPANT FLOW:
Groups:
- Avastin, Radiation, Temozolomide, and Irinotecan: Treatment with standard XRT (radiation) and daily temozolomide 75 mg/m2/day for 6.5 weeks of XRT. Avastin will be administered 10 mg/kg every other week beginning a minimum of 28 days after last major surgical procedure, open biopsy, or significant traumatic injury.
  Following completion of XRT, patients will receive 6 cycles of Avastin, temozolomide, and irinotecan. Beginning a minimum of 14 days after last XRT, Avastin at 10 mg/kg with irinotecan every other week; temozolomide will be given at 200 mg/m2/day on the 1st 5 days of each 28-day cycle. The irinotecan dose will depend on whether the patient is taking enzyme-inducing antiepileptic drugs (EIAED). (EIAED:340 mg/m2 every other week, non-EIAED:125 mg/m2.)
Period: Overall Study
Arm/Group | Avastin, Radiation, Temozolomide, and Irinotecan
Started | 125
Completed | 125
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Avastin, Radiation, Temozolomide, and Irinotecan
Number analyzed (Participants) | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 74

OUTCOME MEASURES:

1. Primary Outcome: 16-month Overall Survival (OS)
Description: Percentage of participants surviving sixteen months from the start of study treatment. OS was defined as the time from the date of study treatment initiation to the date of death due to any cause.
Time Frame: 16 months
Population: Intent to treat
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Avastin, Radiation, Temozolomide, and Irinotecan
Number analyzed (Participants) | 125
percentage of participants | 64.8 [55.7 to 72.5]

2. Secondary Outcome: 12-month Progression-free Survival (PFS)
Description: Percentage of participants surviving twelve months from the start of study treatment without progression of disease. PFS was defined as the time from the date of study treatment initiation to the date of the first documented progression according to the Macdonald criteria, or to death due to any cause.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Avastin, Radiation, Temozolomide, and Irinotecan
Number analyzed (Participants) | 125
percentage of participants | 63.2 [54.1 to 71.0]

3. Secondary Outcome: Number of Patients Experiencing a Central Nervous System (CNS) Hemorrhage or a Systemic Hemorrhage
Description: Number of times a CNS hemorrhage or systemic hemorrhage was experienced
Time Frame: 55 months
Measure: Number; unit: participants
Arm/Group | Avastin, Radiation, Temozolomide, and Irinotecan
Number analyzed (Participants) | 125
participants
  Gr.2 Central Nervous System (CNS) Hemorrhage | 1
  Gr.3 Central Nervous System (CNS) Hemorrhage | 0
  Gr.4 Central Nervous System (CNS) Hemorrhage | 1
  Gr.5 Central Nervous System (CNS) Hemorrhage | 0
  Gr.2 Systemic Hemorrhage | 1
  Gr.3 Systemic Hemorrhage | 0
  Gr.4 Systemic Hemorrhage | 0
  Gr.5 Systemic Hemorrhage | 0

4. Secondary Outcome: Number of Patients Experiencing a Grade ≥ 4 Hematologic or Grade ≥ 3 Non-hematologic Toxicity
Description: Number of times a grade ≥ 4 hematologic or grade ≥ 3 non-hematologic toxicity was experienced
Time Frame: 55 months
Measure: Number; unit: participants
Arm/Group | Avastin, Radiation, Temozolomide, and Irinotecan
Number analyzed (Participants) | 125
participants
  Grade ≥ 4 Hematologic Toxicities | 20
  Grade ≥3 Non-hematologic Toxicities | 49

ADVERSE EVENTS:
Time Frame: 55 months
Description: Adverse events collected using Common Terminology Criteria for Adverse Events (CTCAE) v.3.0 and converted to v.4.0 for ClinicalTrials.gov entry.
Arm/Group | Avastin, Radiation, Temozolomide, and Irinotecan
Serious Adverse Events (participants affected / at risk) | 35/125
Other Adverse Events (participants affected / at risk) | 45/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Avastin, Radiation, Temozolomide, and Irinotecan (N=125)
Anemia (Blood and lymphatic system disorders) | 4
Atrial fibrillation (Cardiac disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Death NOS (General disorders) | 2
Fatigue (General disorders) | 1
Sudden death NOS (General disorders) | 1
Bone infection (Infections and infestations) | 1
Infections and infestations - Other, specify (Infections and infestations) | 1
Infections and infestations - Other, specify: Infecti (Infections and infestations) | 2
Lung infection (Infections and infestations) | 3
Skin infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Neutrophil count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 4
White blood cell decreased (Investigations) | 3
Dehydration (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrospinal fluid leakage (Nervous system disorders) | 1
Cognitive disturbance (Nervous system disorders) | 1
Headache (Nervous system disorders) | 2
Intracranial hemorrhage (Nervous system disorders) | 2
Peripheral motor neuropathy (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 13
Confusion (Psychiatric disorders) | 5
Psychosis (Psychiatric disorders) | 1
Thromboembolic event (Vascular disorders) | 7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Avastin, Radiation, Temozolomide, and Irinotecan (N=125)
Fatigue (General disorders) | 10
Neutrophil count decreased (Investigations) | 25
Platelet count decreased (Investigations) | 23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes